CLINICAL TRIAL: NCT01247896
Title: A Phase 1 Placebo-controlled Trial to Assess the Safety, Tolerability, and Pharmacokinetics of Single Escalating Oral Doses of PF-05190457 Under Fasted and Fed Conditions in Healthy Adult Subjects
Brief Title: Single Dose Escalation Study of PF-05190457 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3301001
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-5190457

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: PF-05190457
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05190457 — Single Dose 2 mg
  Arms: Active
Drug: PF-05190457 — Single Dose 10 mg
  Arms: Active
Drug: PF-05190457 — Single Dose 30 mg
  Arms: Active
Drug: PF-05190457 — Single Dose 100 mg
  Arms: Active
Drug: PF-05190457 — Single Dose 300 mg
  Arms: Active
Drug: PF-05190457 — Single Dose 600 mg
  Arms: Active
Drug: PF-05190457 — Single Dose - to be determined with food
  Arms: Active
Drug: PF-05190457 — Single Dose - to be determined
  Arms: Active
Drug: Placebo — Single Dose Placebo
  Arms: Placebo

SUMMARY:
PF-05190457 is a novel compound proposed for the treatment of Type 2 diabetes mellitus. The purpose of the study is to evaluate the safety and tolerability of PF-05190457 after administration of a single dose to healthy volunteers and to evaluate the plasma drug concentrations after single dose in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females (non-childbearing) between the ages of 18 and 55 with BMI of 17.5 to 30.5 kg/m2; and a total body weight between 50 kg (110 lbs) and 100 kg (220 lb) inclusive

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PF-05190457 will be assessed by physical examinations, adverse event monitoring, 12-lead ECGs, continuous cardiac monitoring over the first 8 hours after dosing, vital sign and clinical safety laboratory measurements | 8 weeks
The single dose PK of PF-05190457 will be described by estimating parameters of AUC(0-infinity), AUC(0-last), AUC(0-24), Cmax, Tmax, CL/F, Vz/F and half-life (t1/2), as the data permit | 48 hour

SECONDARY OUTCOMES:
PK of PF-05190457 in the fed condition will be described by estimating parameters of AUC(0-infinity), AUC(0-last), AUC(0-24), Cmax, Tmax, CL/F, Vz/F and half-life (t1/2), | 48 hour
Gastric half-emptying time (GET½), the duration of the lag phase (Tlag), gastric emptying coefficient (GEC) | Day 1 for Periods 1 and 2, for Cohort 3.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Cobbina E, Lee MR, Leggio L, Akhlaghi F. A Population Pharmacokinetic Analysis of PF-5190457, a Novel Ghrelin Receptor Inverse Agonist in Healthy Volunteers and in Heavy Alcohol Drinkers. Clin Pharmacokinet. 2021 Apr;60(4):471-484. doi: 10.1007/s40262-020-00942-7. Epub 2020 Nov 5. PMID 33155163
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3301001&StudyName=Single%20Dose%20Escalation%20Study%20of%20PF-05190457%20in%20Healthy%20Volunteers